CLINICAL TRIAL: NCT01698944
Title: Cardiovascular Effects on Growth Hormone Replacement Therapy in Adults With Primary or Secondary Childhood Onset Growth Hormone Deficiency
Brief Title: Cardiovascular Effects on Growth Hormone Therapy in Adults With Growth Hormone Deficiency
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was prematurely terminated due to low recruitment
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHDADULT-1112
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somatropin (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Initial dose 0.5 IU/day and escalated up to maximum dose the first 6 months. Maximum dose 3.0 IU/day for 18 months. Injected subcutaneously (s.c., under the skin) daily

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the effect of growth hormone on left ventricle morphology and function (systolic and diastolic).

ELIGIBILITY:
Inclusion Criteria:

* Adult growth hormone deficiency
* At least 2 years without growth hormone treatment

Exclusion Criteria:

* Supine blood pressure above 160 mmHg systolic or above 100 mmHg diastolic
* Pregnancy

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2001-05-16 (Actual); Primary Completion 2002-11-18 (Actual); Study Completion 2002-11-18 (Actual)

PRIMARY OUTCOMES:
Left Ventricular systolic function
Left Ventricular diastolic function

SECONDARY OUTCOMES:
Body composition
Fasting glucose
HbA1c (glycosylated haemoglobin)
Oral glucose tolerance test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Athens, Greece

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com